CLINICAL TRIAL: NCT05204069
Title: Screening for 3-D Visual Disorders in Preschool Children, VISION Study
Brief Title: Screening for 3-D Visual Disorders in Preschool Children
Acronym: VISION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP201100; 2019-A03128-49 (Registry Identifier: ANSM)
Record Dates: First submitted 2021-09-22; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-09

CONDITIONS: Amblyopia; Strabismus; Anisometropia
MeSH Terms: conditions — Amblyopia; Strabismus; Anisometropia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three-dimensional screening for visual disorders using the RetinoMax Device (Experimental): Instillation of cyclopentolate of 3 drops of cyclopentolate at T0',T5' and t10' with to induce a certain level of cycloplegia and evaluate manifest refraction at t45' using the RetinoMax Device.
  Interventions: Drug: Instillation of cyclopentolate
- Non-standardized device for usual vision disorders (Active Comparator): Screening device for usual vision disorders, performed by the school doctor during the usual prevention visit, with the tools used in the school doctor's current practice, non-standardized, according to his preference
  Interventions: Drug: Instillation of cyclopentolate

INTERVENTIONS:
Drug: Instillation of cyclopentolate — Instillation of cyclopentolate of 3 drops of cyclopentolate at t0',t5' and t10' with to induce a certain level of cycloplegia and evaluate manifest refraction at t45' using the RetinoMax Device.

SUMMARY:
Visual screening is necessary among pre-school children as they found themselves in a critical period of visual developement. To date, there are no national vision screening program that has been implemented nationwide. Vision is a pilot feasibility multicentric cluster study comparing the sensitivity of "AFSOP 3 dimensional visual screening protocol in a population of 3 to 4-year-old pre-school children conducted in 4 kindergarten preschools in Paris with gold-standard ophthalmic examination confirmation.

DETAILED DESCRIPTION:
Visual screening is necessary among pre-school children as they found themselves in a critical period of visual developement. To date, there are no national vision screening program that has been implemented nationwide. Methodology: The "Association Française de Strabologie et d'Ophtalmologie Pédiatrique" AFSOP proposed criteria based on a 3-dimensions visual screening to assess whether or not a child presents risk factors of amblyopia such as ametropia, strabismus and anisometropia. Vision is a pilot feasibility multicentric cluster study comparing the sensitivity of "AFSOP 3 dimensional visual screening protocol in a population of 3 to 4-year-old pre-school children conducted in 4 kindergarten preschools in Paris with gold-standard ophthalmic examination confirmation. Expected results: We assume that a vision screening operated with the AFSOP 3 dimension screening recommendations and conducted by paramedical actors such as orthoptists will prove more sensitive and easier to implement on a national scale.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 4 years
* Enrolled in kindergarten in the first section
* In the 19th district of Paris
* Who should benefit from visual screening via the school medical service

Exclusion Criteria:

* Children who do not speak French
* Children who are physically or cognitively unable to participate in the screening

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Screening for 3-dimensional visual disorders | 1 day
  Sensitivity of the " AFSOP 3-dimensional screening" vs "PARIS protocol screening" using a comprehensive ophthalmological examination as a gold standard

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel BUI-QUOC, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debre Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided